CLINICAL TRIAL: NCT06444503
Title: Creation of a Biological Collection to Study the Pathophysiology and Identify Predictive Factors for the Evolution of Bone, Calcium and Growth Plate Pathologies
Brief Title: Clinico-biological Collection of Bone, Calcium and Growth Plate Pathologies
Acronym: OSCAR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0214
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Bone Disorder
MeSH Terms: conditions — Bone Diseases | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, other body fluids and tissues biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients suffering from growth plate or bone pathology: As part of their pathology, patients benefit from clinical monitoring and regular blood and urine tests.
  Interventions: Other: Biological samples; Other: Biological

INTERVENTIONS:
Other: Biological samples — Blood and urine will be taken in larger quantity
Other: Biological — Surgical residues may be preserved in the event of surgery carried out as part of the treatment.

SUMMARY:
The aim of this project is to set up a biological and clinical collection of patients with progressive bone, calcium and growth plate pathologies.

This collection will provide a better understanding of the mechanisms involved in growth plate and bone damage in these diseases and identify factors predictive of progression and new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Children (from birth) with growth plate or bone pathology
* Patients affiliated to or benefiting from a social security scheme
* Patients able to receive information about the study and to understand the information form in order to participate in the study. This implies :
* mastery of the French language
* Not being subject to a restriction of rights by the judicial authorities
* Patients or legal representatives having given their consent to participate in the study (expression of non-opposition).

Exclusion Criteria:

* Patients under legal protection (guardianship, curatorship or safeguard of justice)
* Pregnant or breast-feeding women

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with with growth plate or bone pathology.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2034-09-16 (Estimated); Study Completion 2034-09-16 (Estimated)

PRIMARY OUTCOMES:
Building a collection of biological samples and clinical-biological data from patients presenting bone, calcium and growth plate pathologies | Day 0 and through study completion, an average of 5 years
  Blood and urine sampling

SECONDARY OUTCOMES:
Identification of potential markers of disease progression based on new knowledge. | Day 0 and through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas EDOUARD, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Toulouse Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No